CLINICAL TRIAL: NCT00156962
Title: A Randomized, Open-Label Study to Assess the Safety of Epoetin Alfa Manufactured by Deep Tank Technology and Epoetin Alfa Manufactured by Roller Bottle Technology in Subjects With Chronic Kidney Disease Not on Dialysis
Brief Title: Epoetin Alfa (EPO) in Subjects With Chronic Kidney Disease (CKD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Regulatory decision not to proceed
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040259; NOT APPLILCABLE
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Kidney Disease
Keywords: Epogen; Procrit; Chronic Kidney Disease; Anemia Treatment
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Epoetin Alfa

ARMS (2):
- Epoetin alfa RB (Active Comparator)
  Interventions: Drug: Epoetin alfa RB
- Epoetin alfa DT (Experimental)
  Interventions: Drug: Epoetin alfa DT

INTERVENTIONS:
Drug: Epoetin alfa DT — Receive drug at same frequency and dose as at the time of randomization Change dose by+/- 25% in order to maintain Hb between 11.0 - 13.0 g/dL
  Arms: Epoetin alfa DT
Drug: Epoetin alfa RB — Receive drug at same frequency and dose as at the time of randomization Change dose by+/- 25% in order to maintain Hb between 11.0 - 13.0 g/dL
  Arms: Epoetin alfa RB

SUMMARY:
The purpose of this study is to look at subject incidence of adverse events.

DETAILED DESCRIPTION:
To determine whether Epoetin alfa manufactured by a roller bottle technology (Epoetin alfa RB) and Epoetin alfa manufactured by a deep tank process (Epoetin alfa DT) have a comparable safety profile when administered to patients with CKD not on dialysis.

ELIGIBILITY:
Inclusion Criteria: - ≥ 18 years of age - CKD not on dialysis: estimated glomerular filtration rate (GFR) of 15mL/min to 60 mL/min (Modification of Diet in Renal Disease [MDRD] equation) - Clinically stable - Mean of all screening/baseline hemoglobin (Hb) values between 11.0 to 13.0 g/dL - Currently receiving Epoetin alfa RB (ie. Epogen or Procrit) at the same dosing frequency for at least four weeks prior to randomization with no more than 1 missed or withheld dose in each of the 2 week periods - Adequate iron stores (transferrin saturation > 15.0%) - No prior use of erythropoietic agents other than Epogen, Procrit or Aranesp Exclusion Criteria: - Currently receiving treatment with any erythropoietic stimulating protein other than Epogen or Procrit. - Prior use of erythropoietic agents other than Epogen, Procrit or Aranesp. - Uncontrolled hypertension (defined as diastolic blood pressure [BP] > 110 mmHg or systolic BP > 180 mmHg during screening). - Grand mal seizure within the last 6 months prior to screening. - Acute myocardial ischemia; hospitalization for congestive heart failure or myocardial infarction within 12 weeks before randomization. - Stroke (hemorrhagic or ischemic) or transient ischemic attack within 12 weeks before randomization. - Major surgery within 3 months prior to screening (excluding vascular access surgery). - Clinical evidence of systemic infection or inflammatory disease at the time of screening and up until randomization. - Known history of severe hyperparathyroidism (intact parathyroid hormone [iPTH] >1500 pg/ml or bio-intact parathyroid hormone [biPTH] > 800 pg/ml within 3 months prior to randomization). - Known positivity for HIV antibody or hepatitis B surface antigen. - Clinical evidence of current malignancy with the exception of basal cell or squamous cell carcinoma of the skin. - Blood transfusions within 8 weeks prior to screening or active bleeding. - Androgen therapy within 8 weeks prior to screening. - Interferon therapy.

Patients known to have tested positive at any time in the past for antibodies to erythropoietic proteins. - Systemic hematological disease (eg. sickle cell anemia, myelodysplastic syndromes, hematological malignancy); myeloma; hemolytic anemia. - Other investigational products are excluded. - Subject is currently enrolled in, or has not yet completed a period of at least 30 days since ending other investigational device or drug trial(s). - Psychiatric, addictive, or any other disorder that compromises ability to give truly informed consent for participation in this study. - Pregnant or breast feeding (women of child-bearing potential must be taking adequate contraceptive precautions). - Anticipating or scheduled for a living-related kidney transplant. - Currently receiving home hemodialysis treatment. - Currently receiving immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Estimated)
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Subject incidence of adverse events | Entire Study

SECONDARY OUTCOMES:
Epoetin alfa antibodies | Entire Study
Changes from baseline laboratory and vital signs | Entire Study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_05_EPO_20040259.pdf
- See also: FDA-approved Drug Labeling — http://www.epogen.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com